CLINICAL TRIAL: NCT01697228
Title: The Effects of Vitamin D Supplementation on Glycemic Control and Proinflammatory Markers Involved in Microvascular Complications in Adolescents With Type 1 Diabetes.
Brief Title: The Effects of Vitamin D on Glycemic Control and Proinflammatory Markers in Adolescents With T1DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Roshanak Monzavi MD, Assistant Professor, Center for Endocrinology, Diabetes, and Metabolism, Children's Hospital Los Angeles
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 11-00352
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Type 1 Diabetes; Vitamin D Deficiency/Insufficiency
Keywords: Diabetes; Vitamin D; Proinflammatory markers
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Vitamin D Deficiency; Diabetes Mellitus | interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate treatment group (Other): This group will receive vitamin D supplementation for the first 6 months, then will be monitored off vitamin D for the next 6 months.
  Interventions: Dietary Supplement: Vitamin D
- Delayed treatment group (Other): This group will be monitored for the first 6 months, and then will be given vitamin D for the next 6 months.
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D

SUMMARY:
The investigators are conducting a prospective cross-over study to evaluate the effects of vitamin D supplementation on diabetes control and the pro-inflammatory markers involved in microvascular complications in adolescents with Type 1 Diabetes. The investigators expect to see a significant improvement in glycemic control and a reduction of serum pro-inflammatory markers in adolescents with Type 1 Diabetes and vitamin D deficiency or insufficiency, who are treated with vitamin D.

ELIGIBILITY:
Inclusion Criteria:

1. Between 13 to 21 years of age, with at least Tanner stage 4 sexual maturity for males or post-menarchal females, and T1DM for at least 1 year. To ensure that inclusion criteria for sexual maturity are met, a physical exam for research purposes will be performed.
2. HbA1c between 7 to 9%
3. Adequate renal function (serum creatinine < 1.5 mg/dL in males and < 1.2 mg/dL in females) and adequate liver function (AST and ALT < 2.5 times the upper limit of normal)
4. Vitamin D insufficiency or deficiency (25-OH vit D level < 30ng/mL) which will be determined on initial screening labs after consenting subjects.

Exclusion Criteria:

1. Less than 13 or greater than 21 years of age
2. Less than Tanner stage 4 sexual maturity for males or pre-menarche
3. HbA1c less than 7% or greater than 9%
4. T1DM for less than 1 year
5. Vitamin D sufficient (25-OH vit D level > 30 ng/mL)
6. Currently taking any medication that can interfere with vitamin D synthesis or metabolism, including but not limited to Orlistat, Phenobarbital, Dilantin, Anti-tuberculosis drugs
7. Currently taking any medication other than insulin that alters blood glucose levels, including but not limited to systemic glucocorticoids
8. Inadequate renal function (serum creatinine > 1.5mg/dL in males and > 1.2mg/dL in females) or inadequate liver function (AST and ALT > 2.5 times the upper limit of normal)
9. Evidence of malabsorption or short gut.

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | 6 months
  The primary endpoint in this study will be the difference in change in Hemoglobin A1c between the treatment and non-treatment periods (6 months)

SECONDARY OUTCOMES:
Pro-inflammatory markers | 6 months
  Change in pro-inflammatory markers (CRP, IL-6, TNF-α) between treatment and non-treatment periods
Vitamin D level and proinflammatory markers | 6 months
  Correlation between change in vitamin D levels and circulating pro-inflammatory markers, including CRP, IL-6, and TNF-α
Vitamin D levels on insulin requirements | 6 months
  Correlation between the change of vitamin D levels on insulin requirements
Vitamin D level and HbA1c | 6 months
  Correlation between the change in vitamin D level in the blood and change in HbA1c
Baseline differences between vitamin D deficient & sufficient subjects | Baseline
  Comparison of baseline differences between vitamin D deficient/insufficient subjects and vitamin D sufficient subjects (including pro-inflammatory markers, HbA1c and total daily insulin requirements

CONTACTS AND LOCATIONS:
Overall Officials: Roshanak Monzavi, M.D., Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States